CLINICAL TRIAL: NCT02397772
Title: The Impact of Different Treatment Strategies on the Transmission Dynamics of Soil-transmitted Helminths: a Cluster Randomised Trial in Kenya
Brief Title: Impact of Alternative Treatment Strategies and Delivery Systems for Soil-transmitted Helminths in Kenya
Acronym: TUMIKIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Kenya Ministry of Health (Other Government); Imperial College London (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1354; 2826 (Other: Kenya Medical Research Institute Ethics Review Committee)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Helminthiasis; Nematode Infection; Disease Transmission, Infectious
Keywords: Soil-transmitted helminths; Intestinal Nematodes; Hookworm; Ascaris; Mass Treatment; Kenya
MeSH Terms: conditions — Helminthiasis; Nematode Infections; Communicable Diseases; Ancylostomiasis | interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Annual school-based deworming (Active Comparator): Pre-school and school children (typically 2-14 years) will receive albendazole treatment from trained school teachers, as part of the ongoing national school-based deworming programme.
  Interventions: Drug: albendazole
- Annual community-based deworming (Experimental): Standard school-based deworming supplemented by annual community-based deworming (2-99 years). All household members who are not enrolled in school will receive albendazole treatment from trained community health workers.
  Interventions: Drug: albendazole
- Biannual (Experimental): Biannual school- and community-based deworming (2-99 years). All household members who are not enrolled in school will receive albendazole treatment from trained community health workers
  Interventions: Drug: albendazole

INTERVENTIONS:
Drug: albendazole — Single dose of albendazole (400 mg)
  Other Names: Zentel

SUMMARY:
The mainstay of control of soil-transmitted helminths (STH) is school-based deworming but recent modelling has highlights that in all but low very transmission settings, the treatment of school-aged children is unlikely to interrupt transmission, and that new treatment strategies are required. This study seeks to answer the question: is it possible to interrupt the transmission of STH and if so, what is the most cost-effective treatment strategy and delivery system to achieve this goal? In this study, two paired community cluster randomised trials in different settings in Kenya will evaluate the impact and cost-effectiveness of annual school-based deworming, annual community-based deworming, and biannual community-based deworming. The interventions are (i) annual mass anthelmintic treatment delivered either to pre-school and school-aged children, as part of a national school-based deworming programme, or to the entire community delivered by community health workers. The primary outcome measure is the prevalence of hookworm infection (the most common STH species), assessed by periodic cross-sectional, age-stratified parasitological surveys. Secondary outcomes include intensity of hookworm, prevalence and intensity of Ascaris lumbricoides, treatment coverage, and among a randomly selected sub-sample of participants who will be followed longitudinally, worm burden and proportion of eggs unfertilised. A nested process evaluation, using semi-structured interviews, focus group discussions and a stakeholder analysis will investigate the community acceptability, feasibility given the local and regional health system structures and processes, and scale-up of the interventions.

DETAILED DESCRIPTION:
The study will be conducted in two settings of Kenya that have contrasting epidemiological and programmatic characteristics, Kwale County on the south Kenyan coast and Bungoma County in western Kenya. Allocation to study group will be by cluster, using predefined units used in public health provision - termed Community Units (CUs), which comprise approximately 1,000 households or 5,000 people. CUs will be randomized to one of three groups, receiving either (i) annual school-based deworming; (ii) annual community-based deworming; (iii) biannual community-based deworming. In nine CUs, a longitudinal study will be conducted in order to better understand the transmission dynamics of STH.

ELIGIBILITY:
Inclusion Criteria:

* Usual resident of study community or student enrolled in study school;
* Willingness of adult aged 18 years and above or parent/guardian to provide written informed consent;
* Provision of written assent to participate from children aged 8 years and above.

Exclusion Criteria:

* Visitor to household at time of household visits;
* Refusal of informed consent;
* Refusal to assent by children aged 8 years and above.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21761 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of hookworm in community members | Endline survey conducted, approximately 24 months after starting the intervention
  The prevalence of hookworm will be measured in a final age-stratified, community cross-sectional survey, which will be conducted approximately 24 months after the start of the intervention. Selected individuals will be asked to provide a stool sample which will be examined in duplicate and within one hour of preparation using the Kato-Katz method. Parasite prevalence will be defined as the proportion of slides that are positive for hookworm eggs. A baseline survey will be conducted prior to implementing the intervention and an interim survey conducted at 12 months. In a random subset of individuals, additional confirmatory diagnosis of infection will be based on real-time polymerase chain reaction (PCR).

SECONDARY OUTCOMES:
Prevalence of Ascaris lumbricoides in community members | Endline survey conducted, approximately 24 months after starting the intervention
  The prevalence of Ascaris will be measured in a final age-stratified, community cross-sectional survey, which will be conducted approximately 24 months after the start of the intervention. Selected individuals will be asked to provide a stool sample which will be examined in duplicate and within one hour of preparation using the Kato-Katz method. Parasite prevalence will be defined as the proportion of slides that are positive for hookworm eggs. A baseline survey will be conducted prior to implementing the intervention and an interim survey conducted at 12 months. In a random subset of individuals, additional confirmatory diagnosis of infection will be based on real-time PCR.
Intensity of infection for each STH species | Endline survey conducted, approximately 24 months after starting the intervention
  The intensity of STH species will be measured in a final age-stratified, community cross-sectional survey, which will be conducted approximately 24 months after the start of the intervention. Selected individuals will be asked to provide a stool sample which will be examined in duplicate and within one hour of preparation using the Kato-Katz method. Intensity of infection will be quantified as eggs per gram of faeces. A baseline survey will be conducted prior to implementing the intervention and an interim survey conducted at 12 months.
Treatment coverage | Up to month following treatment
  • Treatment coverage will be measured using both routine data, and data collected during scheduled STH stool surveys. Teachers and community health workers (CHWs) will be provided with treatment registers and asked to provide a full record of all individuals who have received treatment. To augment these data, population-based coverage surveys using multistage clustering sampling will be carried out among a random subsample of communities.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Pullan, PhD, Principal Investigator — London School of Hygeiene & Tropical Medicine
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Derived] Halliday KE, Oswald WE, Mcharo C, Beaumont E, Gichuki PM, Kepha S, Witek-McManus SS, Matendechero SH, El-Busaidy H, Muendo R, Chiguzo AN, Cano J, Karanja MW, Musyoka LW, Safari TK, Mutisya LN, Muye IJ, Sidigu MA, Anderson RM, Allen E, Brooker SJ, Mwandawiro CS, Njenga SM, Pullan RL. Community-level epidemiology of soil-transmitted helminths in the context of school-based deworming: Baseline results of a cluster randomised trial on the coast of Kenya. PLoS Negl Trop Dis. 2019 Aug 9;13(8):e0007427. doi: 10.1371/journal.pntd.0007427. eCollection 2019 Aug. PMID 31398204
- [Derived] Pullan RL, Halliday KE, Oswald WE, Mcharo C, Beaumont E, Kepha S, Witek-McManus S, Gichuki PM, Allen E, Drake T, Pitt C, Matendechero SH, Gwayi-Chore MC, Anderson RM, Njenga SM, Brooker SJ, Mwandawiro CS. Effects, equity, and cost of school-based and community-wide treatment strategies for soil-transmitted helminths in Kenya: a cluster-randomised controlled trial. Lancet. 2019 May 18;393(10185):2039-2050. doi: 10.1016/S0140-6736(18)32591-1. Epub 2019 Apr 18. PMID 31006575
- [Derived] Brooker SJ, Mwandawiro CS, Halliday KE, Njenga SM, Mcharo C, Gichuki PM, Wasunna B, Kihara JH, Njomo D, Alusala D, Chiguzo A, Turner HC, Teti C, Gwayi-Chore C, Nikolay B, Truscott JE, Hollingsworth TD, Balabanova D, Griffiths UK, Freeman MC, Allen E, Pullan RL, Anderson RM. Interrupting transmission of soil-transmitted helminths: a study protocol for cluster randomised trials evaluating alternative treatment strategies and delivery systems in Kenya. BMJ Open. 2015 Oct 19;5(10):e008950. doi: 10.1136/bmjopen-2015-008950. PMID 26482774